CLINICAL TRIAL: NCT04175730
Title: Prostate Cancer Detection Using a Quantitative Screening MRI Protocol
Brief Title: Prostate Cancer Detection Screening MRI Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Michael R Abern, Principal Investigator, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2019-0231
Record Dates: First submitted 2019-10-28; First posted 2019-11-25 (Actual); Results first posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: 50 men with clinical suspicion of PCa (elevated Prostate specific antigen (PSA) and/or abnormal DRE) will be enrolled into a prospective protocol and will undergo detection protocol MRI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MRI and Ultrasound (Other): men with elevated PSA or abnormal DRE for which prostate biopsy is indicated and mpMRI positive for suspected prostate cancer followed by MRI/ultrasound fusion directed prostate needle biopsies
  Interventions: Device: Ultrasound and MRI
- Ultrasound (Other): men with elevated PSA or abnormal DRE for which prostate biopsy is indicated and mpMRI negative for suspected prostate cancer followed by standard ultrasound guided prostate needle biospies
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound and MRI — A single subsequent ultrasound guided prostate biopsy with MRI fusion
  Arms: MRI and Ultrasound
Device: Ultrasound — A single subsequent ultrasound guided prostate biopsy
  Arms: Ultrasound

SUMMARY:
Whether a quantitative detection specfic magnetic resonance imaging (MRI) protocol improves prostate cancer (PCa) detection in biopsy naïve men is not adequately studied.

DETAILED DESCRIPTION:
This will be a 2 arm prospective clinical trial. Men with clinical suspicion for PCa but no prior prostate biopsy will be enrolled from the University of Illinois (UI) Health Urology clinics. All eligible men will be screened and enrolled by the clinical research coordinator. Enrolled men will undergo detection protocol MRI at the UIC Advanced Imaging Center (AIC) prior to diagnostic biopsy. The MRI will be processed by the study team and evaluated for areas suspicious for high grade PCa by a board certified clinical radiologist. Subjects with MRI with no suspicious areas for high grade PCa will undergo standard of care (SOC) core transrectal ultrasound (TRUS) biopsy. Subject with MRI suspicious for high grade PCa will have 2-4 biopsies guided toward each suspicious lesion using MRI/TRUS fusion biopsies (maximum of 12 cores). All biopsies will undergo SOC histologic processing and interpretation in pathology. Biopsy results will be communicated to the patients by the Urologist performing the biopsy and all additional management will be SOC. This visit will signify the end of the study

ELIGIBILITY:
Inclusion Criteria:

* Adult men between 18 and 80 years of age
* Suspected PCa as defined by elevated PSA ≥4 ng/mL and ≤20 ng/mL and/or abnormal DRE as determined by a physician
* Ability to provide informed consent

Exclusion Criteria:

* Prior prostate biopsy
* Prior diagnosis of PCa
* MRI incompatible implanted medical devices or foreign bodies
* Rectal anatomy incompatible with TRUS biopsy
* Life expectancy <10 years as determined by the treating urologist

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 48 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Abern, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Hospital and Ambulatory Clinics, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRI and Ultrasound | Ultrasound
Started | 27 | 21
Completed | 27 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRI and Ultrasound | Ultrasound | Total
Number analyzed (Participants) | 27 | 21 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 12 | 30
  >=65 years | 9 | 9 | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [57 to 74] | 63 [57 to 72] | 62 [57 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 27 | 21 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 26 | 16 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 7 | 25
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 21 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Grade or High Grade (Gleason Score 7 or Higher) Prostate Cancer as Measured by Histopathology
Description: Per subject prevalence of any grade or high grade (Gleason score 7 or higher) prostate cancer as measured by histopathology. When looking at cells under the microscope, the doctor assigns a grade between 1-5. 1 means almost normal and 5 means very different from normal. Adding to two most common grades determines the Gleason score. Higher numbers indicate a faster growing cancer
Time Frame: 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | MRI and Ultrasound | Ultrasound
Number analyzed (Participants) | 27 | 21
Participants | 11 | 8

2. Primary Outcome: Number of Biopsy Samples With a Prevalence of High Grade (Gleason 7 or Higher) Prostate Cancer as Measured by Histopathology
Description: Per biopsy sample prevalence of high grade (Gleason 7 or higher) prostate cancer as measured by histopathology. When looking at cells under the microscope, the doctor assigns a grade between 1-5. 1 means almost normal and 5 means very different from normal. Adding to two most common grades determines the Gleason score. Higher numbers indicate a faster growing cancer
Time Frame: 19 months
Measure: Count of Units; unit: Biopsy
Units Other Than Participants: Biopsy
Arm/Group | MRI and Ultrasound | Ultrasound
Number analyzed (Participants) | 27 | 21
Number analyzed (Biopsy) | 151 | 252
Biopsy | 8 | 3

3. Primary Outcome: Number of Participants With PI-RADS 4-5 on MRI
Description: The accuracy of the mpMRI (PI-RADS version 2 score) to accurately characterize Gleason 7 or higher prostate cancer as measured by histopathology. When looking at cells under the microscope, the doctor assigns a grade between 1-5. 1 means almost normal and 5 means very different from normal. Adding to two most common grades determines the Gleason score. Higher numbers indicate a faster growing cancer
Time Frame: 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | MRI and Ultrasound | Ultrasound
Number analyzed (Participants) | 27 | 21
Participants | 23 | 5

4. Primary Outcome: Number of Participants With PI-RADS <4 MRI
Description: as for outcome 3
Time Frame: 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | MRI and Ultrasound | Ultrasound
Number analyzed (Participants) | 27 | 21
Participants | 4 | 16

5. Primary Outcome: Number of Participants That Had Adverse Events
Description: Adverse events of prostate biopsy using the Clavien-Dindo scale
Time Frame: 19 months
Measure: Count of Participants; unit: Participants
Arm/Group | MRI and Ultrasound | Ultrasound
Number analyzed (Participants) | 27 | 21
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 19 months
Arm/Group | MRI and Ultrasound | Ultrasound
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/21
Other Adverse Events (participants affected / at risk) | 0/27 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT04175730/Prot_SAP_000.pdf